CLINICAL TRIAL: NCT06310941
Title: Aspiration of Bronchial Secretions With Mechanical Insufflation-Exsufflation and Hypertonic Saline in Bacterial Nosocomial Tracheobronchitis and Pneumonia in Intubated Patients.
Brief Title: Mechanical Insufflation-exsufflation and Hypertonic Saline in Nosocomial Bacterial Respiratory Tract Infection
Acronym: ABSENTA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: FUNDACION PARA LA INVESTIGACION HOSPITAL CLINICO SAN CARLOS (Other)
Responsible Party: Principal Investigator, Miguel Sanchez Garcia, Emeritus Critical Care Department, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABSENTA; Pending (Other: Ceim HCSC (ERB of Hospital Clinico San Carlos)))
Record Dates: First submitted 2024-02-27; First posted 2024-03-15 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Nosocomial Infection; Nosocomial Pneumonia; Tracheobronchitis; Mechanical Ventilation Complication; Endotracheal Intubation
Keywords: mechanical insufflation-exsufflation; cough assist device; hypertonic saline; nosocomial respiratory tract infection; hospital-acquired pneumonia; tracheobronchitis; ventilator-associated pneumonia; nebulization
MeSH Terms: conditions — Cross Infection; Healthcare-Associated Pneumonia; Pneumonia, Ventilator-Associated | interventions — Standard of Care; Saline Solution, Hypertonic; Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: multicenter, randomized, open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard of Care (Active Comparator): Standard of care: Systemic antibiotic therapy according to local protocol and at the discretion of the attending intensivist.
  Interventions: Other: Standard of Care
- Mechanical insufflation-exsufflation with hypertonic saline/hyaluronic acid comination (Experimental): Systemic antibiotic therapy choice according to local protocol and at the discretion of the attending intensivist plus Mechanical insufflation-exsufflation (MI-E sessión tid during the first 48 hours, followed by MI-E if secretions are present or suspected; recommended settings +50 cmH2O/-50 cmH2O) with simultaneous nebulization of hypertonic saline (7%) with hyaluronic acid (0.1%).
  Interventions: Device: Mechanical insufflation-exsufflation; Other: Hypertonic saline with hyaluronic acid
- Mechanical insufflation-exsufflation (Experimental): Systemic antibiotic therapy choice according to local protocol and at the discretion of the attending intensivist plus Mechanical insufflation-exsufflation (MI-E sessión tid during the first 48 hours, followed by MI-E if secretions are present or suspected; recommended settings +50 cmH2O/-50 cmH2O)
  Interventions: Device: Mechanical insufflation-exsufflation

INTERVENTIONS:
Device: Mechanical insufflation-exsufflation — Combined use of mechanical insufflation-exsufflation with nebulized hypertonic saline in intubated patients with nosocomial respiratory tract infection
  Other Names: Cough Assist
  Arms: Mechanical insufflation-exsufflation; Mechanical insufflation-exsufflation with hypertonic saline/hyaluronic acid comination
Other: Standard of Care — systemic antibiotic therapy and catheter suctioning of secretions as recommended by guidelines
  Other Names: Routine care of respiratory tract infection
  Arms: Standard of Care
Other: Hypertonic saline with hyaluronic acid — Commercially available combination of 7% hypertonic saline with 0.1% hyaluronic acid given as nebulization during the MI-E session
  Other Names: (Hyaneb-TM)
  Arms: Mechanical insufflation-exsufflation with hypertonic saline/hyaluronic acid comination

SUMMARY:
Multicenter, randomized open label clinical trial to evaluate IEM and HS as concomitant therapy for respiratory tract infection in patients under artificial ventilation in the ICU.

Lung infection is a serious complication that may occur during hospital stay and may need artificial respiration or even develop during artificial ventilation for other causes.

Current specific treatment consists of intravenous antibiotics. The current study evaluated whether aspiration and drainage of infected sputum helps curing this severe complication and whether nebulized HS has additional benefits, like loosening of secretions, eradicating bacteria or reducing inflammation.

DETAILED DESCRIPTION:
Open label, randomized, multicenter (7 ICUs at 7 hospitals in Spain). The study has 2 main arms, pneumonia and tracheobronchitis.

If the diagnosis is pneumonia, subjects will be randomization to one of 3 study groups:

1. IV Antibiotic therapy
2. IV Antibiotic therapy + mechanical insufflation-Exsugglation (MI-E)
3. IV Antibiotic therapy + MI-E + nebulized hypertonic saline-hyaluronic acid (HS)

If the diagnosis is tracheobronchitis,subjects will be randomization to one of 3 study groups:

1. No specific therapy (recommendation of the Infectious Diseases Society of America)
2. IV Antibiotic therapy (common practice to prevent progressión to pneumona and shorten duration of intubation)
3. MI-E + HS

Safety will be compared by number of adverse events, severe adverse events and mortality between study groups in each main arm. Efficacy will be compared by duration of respiratory support and number of cases with worsening organ dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Nosocomial pneumonia (vHAP or VAP) or nosocomial tracheobronchitis
* Intubated with a cuffed endotracheal tube or tracheostomy cannula.

Exclusion Criteria:

* Ominous prognosis
* Frank hemoptisis
* Barotrauma (pneumothorax or pneumomediastinum)
* Bronchospasm (patients on bronchodilators for previous bronchospasm may be included
* Unstable thoracic cage
* Suspected unmonitored intracraneal hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Median SOFA score increase >2 points on day 4 | inclusion to day 4 after randomization
  Increase in organ dysfunction score from baseline to day 4 after randomization.
Median respiratory support-free days increase at day 28 | Inclusion to day 28 after randomization
  28 minus duration in days on high-flow nasal cannula + invasive ventilation.
Percentage of subjects surviving/dying day 28 | Inclusion to day 28 after randomization
  crude mortality on day 28 after randomization

SECONDARY OUTCOMES:
Subjects with bacterial eradication in respiratory samples at day 4 after randomization | Day 3 to 5 after randomization
  Negative tests for causal microorganism in day 4 samples
Subjects with bacterial eradication in respiratory samples at end of systemic antibiotic therapy | 7 and 14 days after randomization
  Negative culture and molecular test for causative bacteria in samples at end of therapy
Median Length of ICU stay | ICU admission to discharge or death in days
  Duration of ICU stay from admission to discharge or death
Median antibiotic-free days at 28 days | from study inclusion to day 28
  28 minus days without systemic antibiotic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Belén De la Hera Hernanz, PhD, Study Director — Hospial Clinico San Carlos
Locations (8):
- Spain (8):
  - Hospital Vall d´Hebrón., Barcelona, Barcelona
  - Hospital Nuestra Señora de la Candelaria., Santa Cruz de Tenerife, Las Palmas
  - Hospital Clinico San Carlos, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital de la Princesa, Madrid, Madrid
  - Hospital Doce de Octubre, Madrid, Madrid
  - Hospital Álvaro Cunqueiro., Vigo, Pontevedra
  - Virgen de la Salud, Toledo, Toledo

IPD SHARING:
Plan to Share IPD: Yes
Anonymyzed data sheet of all subjects and variables for a pre-specified analysis plan.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After study publication
Access Criteria: Anonymyzed data sheet of all subjects and variables for a pre-specified analysis plan.

REFERENCES:
- [Background] Sanchez-Garcia M, Alvarez-Gonzalez M, Domingo-Marin S, Pino-Ramirez AD, Martinez-Sagasti F, Gonzalez-Arenas P, Cardenal-Sanchez C, Velasco-Lopez E, Nunez-Reiz A. Comparison of Mechanical Insufflation-Exsufflation and Hypertonic Saline and Hyaluronic Acid With Conventional Open Catheter Suctioning in Intubated Patients. Respir Care. 2024 Apr 22;69(5):575-585. doi: 10.4187/respcare.11566. PMID 38307525
- [Background] Ferreira de Camillis ML, Savi A, Goulart Rosa R, Figueiredo M, Wickert R, Borges LGA, Galant L, Teixeira C. Effects of Mechanical Insufflation-Exsufflation on Airway Mucus Clearance Among Mechanically Ventilated ICU Subjects. Respir Care. 2018 Dec;63(12):1471-1477. doi: 10.4187/respcare.06253. Epub 2018 Jul 17. PMID 30018175
- [Background] Knudtzen FC, Sprehn M, Vestbo J, Johansen IS. Mechanical insufflation/exsufflation compared with standard of care in patients with pneumonia: A randomised controlled trial. Eur J Anaesthesiol. 2020 Nov;37(11):1077-1080. doi: 10.1097/EJA.0000000000001209. No abstract available. PMID 33027229
- [Background] Sanchez-Garcia M, Santos P, Rodriguez-Trigo G, Martinez-Sagasti F, Farina-Gonzalez T, Del Pino-Ramirez A, Cardenal-Sanchez C, Busto-Gonzalez B, Requesens-Solera M, Nieto-Cabrera M, Romero-Romero F, Nunez-Reiz A. Preliminary experience on the safety and tolerability of mechanical "insufflation-exsufflation" in subjects with artificial airway. Intensive Care Med Exp. 2018 Apr 3;6(1):8. doi: 10.1186/s40635-018-0173-6. PMID 29616357